CLINICAL TRIAL: NCT03699189
Title: Assessment of ANAIS (Alimentación Normal Con Ajuste de InSulina), a Spanish Version of the DAFNE (Dose Adjustment for Normal Eating) Programme, in Patients With Type 1 Diabetes: a Randomised, Controlled, Parallel Trial
Brief Title: ANAIS, a Spanish Version of the DAFNE Programme
Acronym: ANAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosa María Sánchez Hernández (Other)
Collaborators: Ana M. Wägner (Unknown); Dácil Alvarado-Martel (Unknown); Yaiza López-Plasencia (Unknown); Armando Carrillo-Domínguez (Unknown); Julia Rodríguez-Cordero (Unknown); Francisco J Nóvoa-Mogollón (Unknown); Angelines Jiménez-Rodríguez (Unknown)
Responsible Party: Sponsor-Investigator, Rosa María Sánchez Hernández, Medical Doctor, Hospital Universitario Insular Gran Canaria
Organization: Hospital Universitario Insular Gran Canaria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANAIS
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; education programme; quality of life; dietary freedom; patient empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Participation

STUDY DESIGN:
Intervention Model Description: A randomised, controlled, parallel trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate ANAIS (Experimental): Participants that attend the training course immediately.
  Interventions: Behavioral: Immediate ANAIS
- Delayed ANAIS (No Intervention): Participants that attend the training course a year later.

INTERVENTIONS:
Behavioral: Immediate ANAIS — ANAIS is a structured therapeutic education programme aimed at providing the patients with the necessary skills to manage their diabetes independently and confidently. The programme particularly promotes dietary freedom, in an intensive insulin regime, by enabling effective carbohydrate counting and accurate prandial insulin dose adjustment and avoiding hypoglycaemia.
  ANAIS was organised as a five day (Monday to Friday), seven-hour, outpatient programme using principles of adult education, with explicit learning objectives, in a group setting.
  Arms: Immediate ANAIS

SUMMARY:
ANAIS is a therapeutic education programme for type 1 diabetes based on a flexible insulin regime adjusted to the patient's food intake. Participants are randomised in two groups, to attend the training course immediately (immediate ANAIS) or a year later (delayed ANAIS). The main outcome was HbA1c at one year.

DETAILED DESCRIPTION:
ANAIS (Alimentación Normal con Ajuste de InSulina) is a Spanish version of the DAFNE programme, performed in patients with type 1 diabetes. ANAIS is a randomised, controlled, parallel trial.

ANAIS is a group-based, therapeutic education programme for type 1 diabetes based on a flexible insulin regime adjusted to the patient's food intake.

Participants with type 1 diabetes and an HbA1c between 7 and 10% were recruited from the outpatient clinics in a tertiary care center. They were randomised (opaque, sealed envelopes, 2:1 ratio) to attend the training course immediately (immediate ANAIS) or a year later (delayed ANAIS).

The main outcome was HbA1c at one year. Secondary outcomes included lipids, weight, hypoglycemic events, treatment satisfaction, quality of life and self-defined objectives.

ELIGIBILITY:
Inclusion Criteria:

We considered patients to be eligible if they were aged over 18 years, had type 1 diabetes, had an HbA1c between 7-12%, (or HbA1c < 7% with a history of severe hypoglycemia), duration of diabetes of more than two years without advanced complications and ability to understand written and spoken Spanish.

Exclusion Criteria:

Exclusion criteria included severe psychiatric illness, pregnancy, or other circumstances that, according to the investigators' criteria, could interfere with study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | 1 year
  Glycated hemoglobin

SECONDARY OUTCOMES:
Lipids | Baseline, 3, 6 and 12 month
  Total cholesterol, low density lipoprotein cholesterol, high density lipoprotein and triglycerides (all are expressed in mg/dl)
Weight | Baseline, 3, 6 and 12 month
  weight
Hypoglycemic events | Baseline, 3, 6 and 12 month
  Number of hypoglycemic events
Treatment satisfaction | Baseline, 3, 6 and 12 month
  Degree of treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ). Minimum score 0 points, maximum score 36 points. Higher values represent a better outcome.
Self-defined objectives | Baseline, 3, 6 and 12 month
  Participants were asked to establish a maximum of 3 personal goals they wanted to achieve related to taking part in the programme
The quality of life | Baseline, 3, 6 and 12 month
  Degree of quality of life measured by Spanish version of Jacobson's Diabetes Quality of Life questionnaire (EsDQoL). Minimum score 43 points, maximum score 210 points. Higher values represent a worse outcome.

IPD SHARING:
Plan to Share IPD: No